CLINICAL TRIAL: NCT03089957
Title: Prevention of Ulinastatin on Acute Respiratory Distress Syndrome (ARDS) A Randomized Controlled Trial
Brief Title: Prevention of Ulinastatin on Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Peking University Shenzhen Hospital (Other); Central Hospital of Zi Bo (Unknown); Beijing Anzhen Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Beijing Shijitan Hospital Affiliated to Capital Medical University (Unknown)
Responsible Party: Principal Investigator, Zhu Xi, M.D. Chief physician, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2016-0001
Record Dates: First submitted 2017-03-12; First posted 2017-03-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Acute Respiratory Distress Syndrome; Critical Illness
Keywords: Acute Respiratory Distress Syndrome; Critical Illness; Randomized Controlled Trial; Ulinastatin
MeSH Terms: conditions — Respiratory Distress Syndrome; Critical Illness | interventions — urinastatin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ulinastatin group (Experimental): 200,000 IU ulinastatin will be dissolved in 100 mL of 0.9% normal saline by continuous intravenous infusion for 1h, 3 times per day for 5 days.
  Interventions: Drug: Ulinastatin; Other: Usual care
- Control group (Placebo Comparator): Control group will be in usual care without any intervention.
  Interventions: Other: Usual care

INTERVENTIONS:
Drug: Ulinastatin — 200,000 IU ulinastatin will be dissolved in 100 mL of 0.9% normal saline by continuous intravenous infusion for 1h, 3 times per day for 5 days.
  Arms: Ulinastatin group
Other: Usual care — Usual care in ICU.

SUMMARY:
Since strategies were applied in intensive care medicine, including low tidal volume ventilation, fluid resuscitation, use of antibiotics, restrictive transfusion strategy and bundle of ventilator therapy, the incidence of Acute Respiratory Distress Syndrome (ARDS) has been decreased recent years. However, the mortality of severe ARDS is still higher to 45%. Few medications did were indicated to be effective in working on development of ARDS. Different with other disease, ARDS were difficult to prevent in its later stage like a domino effect. The medication interventions are all used after ARDS was developed, including ulinastatin. The investigators hypothesized that the key point in failure of medication therapy is the delay timing of medication intervention. If given the preventive strategy, such as ulinastatin, the incidence or the severity of ARDS might be decreased. Therefore this is a randomized controlled trial to test the hypothesis of the preventive effect of ulinastatin in ARDS.

This is a multi-center, randomized, double blinded, placebo controlled study.

DETAILED DESCRIPTION:
Since strategies were applied in intensive care medicine, including low tidal volume ventilation, fluid resuscitation, use of antibiotics, restrictive transfusion strategy and bundle of ventilator therapy, the incidence of Acute Respiratory Distress Syndrome (ARDS) has been decreased recent years. However, the mortality of severe ARDS is still higher to 45%. Few medications did were indicated to be effective in working on development of ARDS. Different with other disease, ARDS were difficult to prevent in its later stage like a domino effect. The medication interventions are all used after ARDS was developed, including ulinastatin. The investigators hypothesized that the key point in failure of medication therapy is the delay timing of medication intervention. If given the preventive strategy, such as ulinastatin, the incidence or the severity of ARDS might be decreased.

Ulinastatin is a urinary trypsin inhibitor (UTI) that inhibits various inflammatory proteases has been widely used in China, Japan, and Korea for the treatment of patients with inflammatory disorders, postoperative organs protection, shock, and pancreatitis.

Therefore this is a randomized controlled trial to test the hypothesis of the preventive effect of ulinastatin in ARDS.

This is a multi-center, randomized, double blinded, placebo controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be more than 18 years old
* Patients are expected to living within 72 hours of ICU admission
* Patients' Lung Injury Prediction Score (LIPS) more than 4 and got at least 1 risk factors as below: bacteremia, sepsis or sepsis shock, pneumonia, multiple fractures, pulmonary contusion, aspiration, multiple blood transfusion, severe acute pancreatitis.

Exclusion Criteria: Patients will be excluded when they are

* diagnosed as ARDS
* without written informed consent
* with HIV infection
* with other immunologic deficiency (leukaemia, immune deficiency syndrome, etc)
* with organ transplantation or bone marrow transplantation
* with chronic pulmonary disease (except for Chronic Obstructive Pulmonary Disease (COPD) or asthma)
* with angitis
* with neutropenia (except for secondary to sepsis)
* using granulocyte-macrophage colony-stimulating factor or granulocyte colony-stimulating factor
* using asprin or clopidogrel
* using glucocorticoid
* withdrawing treatment
* treated by Xuebijing, thymosin, or intravenous immunoglobulin 1 month before enrollment
* enrolled in other clinical trials 3 months before enrollment
* being pregnancy
* being lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
The incidence of ARDS | 3 years

SECONDARY OUTCOMES:
The numbers of ARDS patients who meet the criteria for mild, moderate, and severe using the Berlin Definition, separately. | 3 years
  The severity of ARDS will be assessed by the Berlin Definition in mild, moderate and severe ARDs according to oxygenation.
The number of patients who need mechanical ventilation | 3 years
Lengths of mechanical ventilation | 3 years
Lengths of ICU | 3 years
Lengths of stay | 3 years
The incidence of other organ disorders | 3 years
Mortality of 28 days | 0-28 days
Mortality of 60 days | 0-60 days
Total cost in admission | 3 years
Adverse events related to drugs. | 3 years

OTHER OUTCOMES:
Adverse events | 3 years
  Including white blood cell decrease, eosinophils increase, nausea, vomiting, diarrhoea, liver enzymes increase, allergy, adverse events in injection sites and etc.

CONTACTS AND LOCATIONS:
Overall Officials: Xi Zhu, M.D., Principal Investigator — Peking University Third Hospital
Locations (10):
- China (10):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital ,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Chinese Pla General Hospital, Beijing, Beijing Municipality
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The first affiliated hospital of Guangxi Medical University, Nanning, Guangxi
  - CANGZHOU People's Hospital, Cangzhou, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The second hospital of dalian medical university, Dalian, Liaoning
  - Central Hospital of Zi Bo, Zibo, Shandong

IPD SHARING:
Plan to Share IPD: Undecided
All data will be shared with other researchers in papers.

REFERENCES:
- [Background] Jeong CW, Lee CS, Lee SH, Jeung HJ, Kwak SH. Urinary trypsin inhibitor attenuates liver enzyme elevation after liver resection. Korean J Anesthesiol. 2012 Aug;63(2):120-3. doi: 10.4097/kjae.2012.63.2.120. Epub 2012 Aug 14. PMID 22949978
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Levitt JE, Calfee CS, Goldstein BA, Vojnik R, Matthay MA. Early acute lung injury: criteria for identifying lung injury prior to the need for positive pressure ventilation*. Crit Care Med. 2013 Aug;41(8):1929-37. doi: 10.1097/CCM.0b013e31828a3d99. PMID 23782966
- [Background] Wang Z, Beach D, Su L, Zhai R, Christiani DC. A genome-wide expression analysis in blood identifies pre-elafin as a biomarker in ARDS. Am J Respir Cell Mol Biol. 2008 Jun;38(6):724-32. doi: 10.1165/rcmb.2007-0354OC. Epub 2008 Jan 18. PMID 18203972
- [Derived] Wang Z, Tao L, Yan Y, Zhu X. Rationale and design of a prospective, multicentre, randomised, conventional treatment-controlled, parallel-group trial to evaluate the efficacy and safety of ulinastatin in preventing acute respiratory distress syndrome in high-risk patients. BMJ Open. 2019 Mar 7;9(3):e025523. doi: 10.1136/bmjopen-2018-025523. PMID 30850411